CLINICAL TRIAL: NCT07101016
Title: Effect of Local Use of Non-steroidal Anti-inflammatory Agent (Diclofenac Sodium) With and Without Hyaluronidase on Post-surgical Pain and Swelling: A Randomized Clinical Trial
Brief Title: Effect of Local Use of Non-steroidal Anti-inflammatory Agent (Diclofenac Sodium) With and Without Hyaluronidase on Post-surgical Pain and Swelling
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mariam Hesham Mahmoud Abdelfattah Eissa (Other)
Responsible Party: Sponsor-Investigator, Mariam Hesham Mahmoud Abdelfattah Eissa, Principle investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422023572518
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Root End Resection; Periapical Lesion; Single Rooted Teeth
Keywords: Periapical lesion; Single rooted teeth; Post operative pain; Post operative swelling; Root end resection; Hyaluronidase; Diclofenac Sodium
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No medication (No Intervention): Osseous cavity left with no medication after root end resection
- Different types of medications placed in the osseous cavity after root end resection (Experimental): I1: Diclofenac sodium : 1 mL of gel, of 1 mL of 3 mL/75 mg Diclofenac sodium and 1% Carbopol 940 gel base, will be passively placed in the osseous cavity I2: Hyaluronidase : 1 mL of gel, of 1 ampoule (1500 IU) Hyalase powder in 2.5 mL of 0.9% sodium chloride, and 1% Carbopol 940 gel base, will be passively placed in the osseous cavity I3: Diclofenac sodium and Hyaluronidase: 1 mL of gel, of 1 ampoule (1500 IU) Hyalase powder and 1 ampoule (3 mL/75 mg) of Diclofenac sodium, Carbopol 940 gel base, will be passively placed in the osseous cavity
  Interventions: Drug: Diclofenac Sodium Gel

INTERVENTIONS:
Drug: Diclofenac Sodium Gel — I1: Diclofenac sodium : 1 mL of gel, of 1 mL of 3 mL/75 mg Diclofenac sodium and 1% Carbopol 940 gel base, will be passively placed in the osseous cavity I2: Hyaluronidase : 1 mL of gel, of 1 ampoule (1500 IU) Hyalase powder in 2.5 mL of 0.9% sodium chloride, and 1% Carbopol 940 gel base, will be passively placed in the osseous cavity I3: Diclofenac sodium and Hyaluronidase: 1 mL of gel, of 1 ampoule (1500 IU) Hyalase powder and 1 ampoule (3 mL/75 mg) of Diclofenac sodium, Carbopol 940 gel base, will be passively placed in the osseous cavity
  Arms: Different types of medications placed in the osseous cavity after root end resection

SUMMARY:
The goal of this clinical trial is to evaluate whether locally applied diclofenac sodium, with or without hyaluronidase, can reduce post-surgical pain and swelling in adult male and female patients (18 years or older) with asymptomatic single-rooted teeth and periapical lesions (5-10 mm in diameter). The main questions it aims to answer are:

Does local application of diclofenac sodium reduce postoperative pain and swelling compared to no medication?

Does the combination of diclofenac sodium and hyaluronidase offer greater reduction in postoperative pain and swelling than diclofenac sodium alone?

Researchers will compare four groups (diclofenac only, hyaluronidase only, diclofenac + hyaluronidase, and no medicament) to see if the medicated groups experience significantly less pain and swelling after periapical surgery compared to the control group.

Participants will:

Undergo root canal treatment followed by periapical surgery in a single visit.

Receive a randomly assigned intra-osseous gel (diclofenac, hyaluronidase, both, or none) placed into the surgical cavity.

Record their postoperative pain using a visual analogue scale at specified intervals (6, 12, 24, 48 hours, and 7 days).

Return for clinical assessments of swelling at 24, 72 hours, and 5 days post-surgery

DETAILED DESCRIPTION:
A) Participants, interventions & outcomes 9. Study settings: The study will be carried out in the endodontic clinic at the faculty of dentistry, Cairo University, Cairo governorate, Egypt.

* The dental Unit is ADEC 200 USA.
* The X-ray machine is FONA XDC, Italy.
* The X-ray sensor plate: Digora intraoral digital sensor plate, Soredex, USA.
* The operator is a PhD student in the department of Endodontics.
* Time: 2025 10. Eligibility criteria:

Inclusion criteria:

1. Patients in good physical health; American Society of Anesthesiologists (ASA) class I or II, with no known allergic manifestations to the drugs used in the study and no involvement with other medication during the study (Appendix 2).
2. Patients who are 18 years of age or older, without underlying chronic systemic conditions.
3. Male and female patients.
4. Patients having asymptomatic single rooted teeth with periapical lesions 5-10mm in diameter (Appendix 3).
5. Patients who can understand the visual analogue scale (Appendix 4).
6. Patients who accept to participate in the trial and can sign the informed consent (Appendix 1).

Exclusion criteria

1. Teeth with pathosis associated with vertical root fractures, teeth with coronal perforations, and periodontal pockets (7 mm).
2. Miller class III/IV mobility, compromised crown-to-root ratio, combined endodontic-periodontic lesions
3. Systemic medical diseases and autoimmune diseases
4. Pregnant females
5. Patients allergic to Diclofenac or Hyaluronidase
6. Teeth with previous root canal therapy

11. Interventions Diagnosis The following diagnostic information will be collected to confirm the eligibility of the participants and will be reported in their diagnostic charts (Appendices 2,3)

1. Personal data: only patients who are 18 years or older will be included in the trial.
2. Medical and dental history: only patients with ASA class I or II will be included in the trial.
3. Findings of clinical examination: asymptomatic single rooted teeth, requiring root canal treatment.
4. Findings of radiographic examination: patients with periapical radiolucency ranging from 5-10mm in diameter will be included in the trial. After complete diagnosis, healthy adult patients with a periapical radiolucency 5-10mm in diameter related to asymptomatic single rooted teeth, with no known allergic manifestations to the drugs will be included.

Treatment procedure:

All patients will sign an informed consent form after the surgical and experimental procedures are explained verbally and in writing. Patients will be instructed to use Chlorhexidine Gluconate (0.2%) mouthwash, 10 mL twice daily, 3 days preoperatively.

Root canal procedure: local anesthesia will be administered: infiltration injection of 4% articaine with 1:100000 epinephrine.

Access cavity preparation: will be done, under rubber dam isolation, using a round bur and a tapered stone with round end.

Working length determination: will be established using an apex locator and confirmed with a periapical radiograph, ensuring it is 0.5 mm short of the radiographic apex.

Cleaning and shaping: all patients will receive the same hybrid technique treatment, combining coronal and apical preparations. Coronal shaping will be performed using a crown-down approach with rotary nickel-titanium instruments , while apical preparation will be done manually up to size #45 K-file .

Irrigation protocol: during instrumentation, canals will be irrigated with 1 ml of 2.5% sodium hypochlorite between each file, using a 27-gauge slotted, side-vented needle . Apical patency will be maintained using a #10 K-file throughout the procedure. For the final rinse, 5 ml of 2.5% sodium hypochlorite will be followed by 10 ml of distilled water.

Obturation: drying of the canals will be done using paper points matching the final apical file size. A radiograph will be obtained to ensure proper master cone extension (size 45, taper 0.02) The canals will then be obturated with the cold lateral condensation technique using gutta-percha and a resin-based sealer .

Final restoration: the access cavity will be restored with composite resin .

Surgical procedure:

The surgical procedure will follow the root canal treatment in the same visit.

1. Chlorhexidine Gluconate 4% scrub, will be applied to the surgical site and the surrounding facial area with sterile gauze and left for 1-2 minutes, then rinsed with sterile saline.
2. Supplemental local anesthesia will be administered: infiltration injection of 4% articaine with 1:100000 epinephrine.
3. A submarginal incision will be made near the mucogingival junction using a surgical scalpel blade 15c, extending mesially and distally from the treated tooth.
4. A full thickness mucoperiosteal flap will be raised with a 9 molt mucoperiosteal elevator. The flap will be mobilized, reflected, and carefully retracted during the root-end management. After flap reflection, a minnesota retractor will be positioned on the exposed cortical bone, with light but firm pressure acting as a passive mechanical barrier to the reflected tissues. The flap will be frequently irrigated with sterile saline to prevent dehydration of the periosteal surface.
5. Impact air-handpiece with a tungsten carbide surgical bur will be used for bone cutting.
6. Periapical lesions will be removed with sharp bone curettes and angled periodontal curettes. Root apex will be removed 3 mm perpendicular to the long axis of the root apex (apicectomy) at a 90° angle. Ultrasonic tips will be used for root-end preparation and MTA for the root-end filling material.
7. The patient will be assigned to either group 1 ,group 2, group 3 or group 4 according to the random sequence for the injected medicament as follows:

(1) Diclofenac sodium: 1 mL of gel prepared by incorporating 1 mL of 3 mL/75 mg Voltaren into a 1% Carbopol 940 gel base, will be passively placed in the osseous cavity, (2) Hyaluronidase: 1 mL of gel prepared by dissolving the contents of 1 ampoule (1500 IU) Hyalase powder in 2.5 mL of 0.9% sodium chloride, and then incorporating 1 mL of this solution into a 1% Carbopol 940 gel base, will be passively placed in the osseous cavity, (3) Diclofenac sodium and Hylauronidase: 1 mL of gel prepared by dissolving the contents of 1 ampoule (1500 IU) Hyalase powder directly in 1 ampoule (3 mL/75 mg) of Voltaren (diclofenac sodium), and then incorporating the entire solution into a Carbopol 940 gel base, will be passively placed in the osseous cavity, (4) The osseous cavity will be irrigated with 5ml of 0.9% sodium chloride, to improve postoperative pain and swelling. All solutions will be injected using a 5ml, 21 gauge needle, syringe.

8. All the flaps will be repositioned and sutured with 5-0 nylon non-resorbable interrupted simple sutures, and removed after 7 days.

Soft and hard tissue management will be performed under a surgical microscope (magnification range between 8X and 20X).

Patients will be instructed to continue to use Chlorhexidine Gluconate 0.2% mouthwash, 10 mL twice daily, for an additional 7 days postoperatively beginning 1 day after surgical procedure.

Self-assessment questionnaires will be distributed postoperatively, which will be verbally reviewed by telephone after 6,12, 24, and 48 hours, as well as 7 days after procedure. Patients will also be asked to come back after 24, 72 hours and 5 days to assess the degree of swelling.

Interventions Each osseous cavity will receive 1cc of the injected medication, after root canal preparation, apicectomy, curettage of the lesion and retrofilling with MTA.

Group 1: Diclofenac sodium : 1 mL of gel, of 1 mL of 3 mL/75 mg Diclofenac sodium and 1% Carbopol 940 gel base, will be passively placed in the osseous cavity Group 2: Hyaluronidase : 1 mL of gel, of 1 ampoule (1500 IU) Hyalase powder in 2.5 mL of 0.9% sodium chloride, and 1% Carbopol 940 gel base, will be passively placed in the osseous cavity Group 3: Diclofenac sodium and Hyaluronidase: 1 mL of gel, of 1 ampoule (1500 IU) Hyalase powder and 1 ampoule (3 mL/75 mg) of Diclofenac sodium, Carbopol 940 gel base, will be passively placed in the osseous cavity Group 4: Suturing of the flap with no medicament

Patients will be given a coded sealed packet preoperatively, that contains 1 of the 4 interventions and the following instructions: (1) No medication; (2) Diclofenac sodium; or (3) Hyaluronidase, or (4) Diclofenac sodium and Hyaluronidase. A dental assistant who is unaware of the experimental protocol will place the coded packets.

12. Outcomes: Primary outcome

Postoperative pain intensity measured at 6,12,24, 72 hours and 1 week post-surgical procedure:

Each patient will receive a pain chart containing a 10-cm visual analogue scale (VAS), one for each time interval. The patient will be instructed to rate his/her pain level at the corresponding time interval on a 10-cm visual analogue scale (VAS), scored between 0 (no pain) and 10 (the most unbearable pain). Metin et al. (2018)

Secondary outcome:

Postoperative swelling Each patient will be asked to return for assessment of the swelling, after 24,72 hours and 5 days, which will be conducted by the operator and co-supervisor by comparing the patients initial photograph. The operator and co-supervisor will rate the swelling level at the corresponding time interval as mild (slight puffiness of gum, cheek, or chin but face not distorted), moderate (cheek or chin or both are visibly distorted), and severe (gross distortion of involved part). Morse et al., (1987), Silva et al.(2022)

Tool Unit Time Post-surgical pain Visual analogue scale (VAS) Metin et al. (2018) Categorical 6,12,24,48 hours and 7 days postoperatively Post-surgical swelling Verbal rating scale (VRS) Silva et al.(2022) Categorical 24,72 hours and 5 days postoperatively

13. Participant timeline

Before Endodontic and surgical treatment:

* Patients will be carefully diagnosed; clinician will ensure that they met all the eligibility inclusion criteria, and if eligible, they will be treated over a single visit.
* Patients will be instructed on how to use the pain scale chart (VAS)

During Endodontic and surgical treatment:

* Informed consent will be obtained.
* Patients will undergo root canal therapy
* Patients will then be assigned to one of the four groups of the study, according to the random sequence conducted by the assistant supervisor.
* Surgical intervention will be carried out, following instructions of the assigned group.

After Endodontic and surgical treatment:

* Patients will be instructed to record their pain levels every 6, 12, 24, 48 hours and 7 days according to the given instructions. And swelling will be assessed by the operator and co-supervisor every 24,72 hours and 5 days post-surgical treatment
* Another appointment will be scheduled after 7 days to collect the NRS scores and assess the outcome of the treatment and remove the sutures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in good physical health; American Society of Anesthesiologists (ASA) class I or II, with no known allergic manifestations to the drugs used in the study and no involvement with other medication during the study (Appendix 2).
2. Patients who are 18 years of age or older, without underlying chronic systemic conditions.
3. Male and female patients.
4. Patients having asymptomatic single rooted teeth with periapical lesions 5-10mm in diameter (Appendix 3).
5. Patients who can understand the visual analogue scale (Appendix 4).
6. Patients who accept to participate in the trial and can sign the informed consent (Appendix 1).

Exclusion Criteria:

* 1. Teeth with pathosis associated with vertical root fractures, teeth with coronal perforations, and periodontal pockets (7 mm).

  2. Miller class III/IV mobility, compromised crown-to-root ratio, combined endodontic-periodontic lesions 3. Systemic medical diseases and autoimmune diseases 4. Pregnant females 5. Patients allergic to Diclofenac or Hyaluronidase 6. Teeth with previous root canal therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity | 6,12,24, 72 hours and 1 week post-surgical procedure
  Postoperative pain intensity measured at 6,12,24, 72 hours and 1 week post-surgical procedure:
  Each patient will receive a pain chart containing a 10-cm visual analogue scale (VAS), one for each time interval. The patient will be instructed to rate his/her pain level at the corresponding time interval on a 10-cm visual analogue scale (VAS), scored between 0 (no pain) and 10 (the most unbearable pain). Metin et al. (2018)

SECONDARY OUTCOMES:
Postoperative swelling | 24,72 hours and 5 days
  Each patient will be asked to return for assessment of the swelling, after 24,72 hours and 5 days, which will be conducted by the operator and co-supervisor by comparing the patients initial photograph. The operator and co-supervisor will rate the swelling level at the corresponding time interval as mild (slight puffiness of gum, cheek, or chin but face not distorted), moderate (cheek or chin or both are visibly distorted), and severe (gross distortion of involved part). Morse et al., (1987), Silva et al.(2022)

IPD SHARING:
Plan to Share IPD: No